CLINICAL TRIAL: NCT03596281
Title: An Open-label Phase 1 of Pembrolizumab in Combination with Bevacizumab and Pegylated Liposomal Doxorubicin in Patients with Platinum Resistant Epithelial Ovarian Cancer
Brief Title: Pembrolizumab in Combination with Bevacizumab and Pegylated Liposomal Doxorubicin in Patients with Ovarian Cancer
Acronym: PEMBOV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004197-34; 2016/2456 (Other: CSET number)
Record Dates: First submitted 2018-06-15; First posted 2018-07-23 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Bevacizumab; liposomal doxorubicin

STUDY DESIGN:
Intervention Model Description: Cohort A and B will be opened for inclusions at the same time. Once safety of the dual combinations confirmed in cohorts A and B, cohort C will be opened for inclusions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: pegylated liposomal doxorubicin (PLD)
- Cohort B (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200mg Q3W IV
Drug: Bevacizumab — 400 or 300 mg Q3W IV
  Arms: Cohort B
Drug: pegylated liposomal doxorubicin (PLD) — 15 or 20 or 30 mg/m² Q3W IV
  Arms: Cohort A

SUMMARY:
French multicenter, open-label, phase 1b, evaluating via the mTPI design the paired treatment of pembrolizumab and PLD (cohort A), pembrolizumab and bevacizumab (cohort B) and finally the combination treatment of the three drugs PLD plus bevacizumab and pembrolizumab (cohort C). Thanks to an expansion cohort C+ the ORR will be evaluated in a total of 19 patients at the RP2 D using an exact binomial one-step Fleming-type design.

Cohort A and B will be opened for inclusions at the same time. Once safety of the dual combinations confirmed in cohorts A and B,cohort C will be opened for inclusions.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial and to comply with study visits and procedures as per protocol.
2. Be over 18 years of age on day of signing informed consent.
3. Histologically confirmed diagnosis of epithelial ovarian carcinoma or fallopian tube carcinoma or primary peritoneal carcinoma.
4. Have received a front line platinum-based regimen (administered via either IV or IP route) per local standard of care (SOC) or treatment guideline following the primary or interval debulking surgery with documented disease recurrence.

   Note: Maintenance treatment following the front line treatment is permitted and counted together as part of the front line treatment. The absence of debulking for inoperable patients is permitted.
5. Have fulfilled the following additional requirements regarding prior treatments for recurrent ovarian cancer (ROC). Have received 0 to unlimited additional prior lines for treating ROC and must have a platinum-free interval (PFI) of ≤ 6 months if the last regimen received is a platinum-based.

   Note: PFI is defined as the time elapsed between the last dose of platinum and the documented evidence of disease progression per RECIST 1.1.
6. Prior therapy containing bevacizumab or other vascular endothelial growth factor (VEGF) pathway-target therapy is permitted.
7. HMeasurable disease (RECIST version 1.1) by investigator assessment with at least 1 unidimensional measurable lesion
8. At least one lesion amenable to biopsy, visible by imaging or without radiological guidance (e.g. vaginal lesion
9. Have no evidence or history of gastro-intestinal events defined as grade≥2, perforation, fistula, necrosis, hemorrhage or intraabdominal abscess.
10. Have no history or previous treatment of inflammatory bowel disease.
11. Left ventricular ejection fraction (LVEF) ≥ 50% as determined by gated cardiac radionucleotide scan (MUGA) or echocardiogram. Normal blood pressure (BP) or adequately treated and controlled hypertension (either systolic BP ≤ 140 mmHg and diastolic BP ≤ 90 mmHg). No clinically significant (i.e. active) cardiovascular disease, including: myocardial infarction or unstable angina within ≤ 6 months of inclusion; New York Heart Association (NYHA) ≥grade2 Congestive Heart Failure; poorly controlled cardiac arrhythmia despite medication; peripheral vascular disease grade

    ≥grade3.
12. Have provided tissue from an archival tissue sample if available (i.e. initial debulking or biopsy).
13. Eastern Cooperative Oncology Group (ECOG)- performance status 0-1.
14. Life expectancy ≥ 12 weeks
15. Demonstrate adequate organ function as defined in Table 2, all screening labs should be performed within 10 days of treatment initiation.
16. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
17. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication (Reference Section 5.9.2).

    Subjects of childbearing potential are those who have not been surgically sterilized (hysterectomy, bilateral oophorectomy or bilateral salpingectomy) or have not been free from menses for > 1 year.
18. Patient affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

1. Platinum refractory cancers, defined as lack of response to salvage treatment with a disease recurrence during the first line platinum-based chemotherapy.
2. Patients with PLD-resistant EOC, as evidenced by lack of response or progression within 6 months of the last dose of PLD.
3. Administration of other simultaneous chemotherapy drugs, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period.
4. Has had prior chemotherapy, targeted therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
5. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study treatment.
6. Major surgery within 30 days or bowel resection at cytoreductive surgery within 6 months before the initiation of study treatment.
7. Non-healing wound or significant traumatic injury within 30 days before the initiation of study treatment.
8. Any previous radiotherapy to the abdomen or pelvis.
9. Previous Cerebro-Vascular Accident, Transient Ischaemic Attack or Sub-Arachnoid Haemorrhage.
10. History or evidence of thrombotic or hemorrhagic disorders within 6 months prior to inclusion, and known inherited (genetic) predisposition to thrombosis (such as deficit in protein C/S) or acquired predisposition to thrombosis (such as anti-phospholipid syndromes)
11. Prior history of hypertensive crisis or hypertensive encephalopathy.
12. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
13. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy within 2 years prior to inclusion.
14. Has known symptomatic active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
15. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
16. Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active pneumonitis.
17. Has an active infection requiring systemic therapy.
18. Has a Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the pre-screening or screening visit through 6 months after the last dose of trial treatment
22. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti- PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
23. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
24. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
25. Patient under guardianship or deprived of his liberty by a judicial or administrative decision
26. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective ethic approval (by chair or designee) is given allowing exception to this criterion for a specific subject.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 3 weeks
  For all the cohorts, the dose limiting toxicity (DLT) period to determine the Maximum dose tolerated (MTD) will be 3 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No